CLINICAL TRIAL: NCT00622037
Title: Bilateral, Masked Comparison of PEG-400 Based Artificial Tear and Systane for the Treatment of Dry Eye Signs, Symptoms and Visual Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Dr. Barry Schechter, Florida Microsurgical Eye Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5338
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): PEG-400 based artificial tear
  Interventions: Drug: PEG-400 based artificial tear
- 2 (Active Comparator): Systane
  Interventions: Drug: Systane

INTERVENTIONS:
Drug: PEG-400 based artificial tear — Instill one drop in the randomized eye four times daily. Can be used more frequently if needed
  Arms: 1
Drug: Systane — Instill one drop in the randomized eye four times daily. Can be used more frequently if needed
  Arms: 2

SUMMARY:
To evaluate and compare the effects of PEG-400 based artificial tear and Systane tears in mild-moderate dry eye patients. TBUT, Visual impact and subjective evaluations will be assessed in this month long trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient reported dry eye symptoms (episodic, annoying, activity limiting), SES OD.
* Physician assessment of mild-moderate dry eye
* Patient willing to instill drops QID and complete entire length of protocol.
* TBUT < 10 seconds
* BCVA of 20/30 or better

Exclusion Criteria:

* Current topical cyclosporine use (Restasis)
* Current Systane use
* Refractive surgery within the last 6 months
* Oral or topical corticosteroid use
* Severe dry eye patients by physician assessment
* current active Blepharitis
* Oral Doxycyclines use
* Oral Antihistamine use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Dry Eye Signs | 4 months

SECONDARY OUTCOMES:
Visual Quality | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Schechter, MD, Principal Investigator — Florida Microsurgical Eye Institute
Locations (1):
- Florida Microsurgical Eye Institute, Boynton Beach, Florida, United States